CLINICAL TRIAL: NCT01939418
Title: A Phase Ib Trial of Gemcitabine and Cisplatin With RAD001 in Patients With Metastatic Triple Negative Breast Cancer Proceeding to an Open Label Randomized Phase II Trial Comparing Gemcitabine/Cisplatin With or Without RAD001.
Brief Title: Phase Ib/II Trials of RAD001 in Triple Negative Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, In Hae Park, Principal Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-13-670; 12491 (Other: Korea Food and Drug Administration)
Record Dates: First submitted 2013-08-28; First posted 2013-09-11 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; triple negative breast cancer; gemcitabine; RAD001
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Everolimus; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 (Experimental): gemcitabine 800mg/m2, D1 and D8 iv. every 3 weeks. cisplatin 30mg/m2, D1 and D8 iv. every 3 weeks. RAD001 5mg QD. po.
  Interventions: Drug: RAD001; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: RAD001 — Afinitor 5mg qd. po.
  Other Names: Afinitor; everolimus
Drug: Gemcitabine — gemcitabine 800mg/m2 iv. D1 and D8 every 3 weeks
Drug: Cisplatin — cisplatin 30mg/m2 iv. D1 and D8 every 3 weeks

SUMMARY:
This study consists of two parts. In a phase Ib part, investigators will explore the recommended dose of gemcitabine, cisplatin, and RAD001 combination in patients with metastatic TNBC. After completing the phase Ib part, investigators will review the data and discuss with Novartis before the start of a phase II part. In the phase II part, investigators will compare the efficacy of the gemcitabine and cisplatin with or without RAD001 in patients with metastatic TNBC.

DETAILED DESCRIPTION:
PIK3CA active mutations are the most frequent genetic event in breast cancer, including in TNBC which presents activated PI3K/AKT signaling due to PIK3CA mutation or PTEN deficiency. TNBC cell lines having activated PI3K/AKT signaling showed a high sensitivity to PI3K/mTOR inhibitors. RAD001 is a potent mTOR complex 1 inhibitor and showed to enhance cisplatin or gemcitabine induced apoptosis by inhibiting p53 induced p21 expression.

This study consists of two parts. In a phase Ib part, investigators will explore the recommended dose of gemcitabine, cisplatin, and RAD001 combination in patients with metastatic TNBC. After completing the phase Ib part, investigators will review the data and discuss with Novartis before the start of a phase II part. In the phase II part, investigators will compare the efficacy of the gemcitabine and cisplatin with or without RAD001 in patients with metastatic TNBC.

ELIGIBILITY:
Inclusion Criteria:

* Females with histologically confirmed, metastatic or stage IV breast cancer
* ER/PgR negative or poor (Allred score ≤ 3/8) and HER2 negative breast cancer
* ECOG performance status 0-2
* Age ≥ 20 years
* Previously treated by anthracycline and taxane in adjuvant/neoadjuvant or metastatic setting
* ≤ 2 chemotherapy regimens for metastatic disease
* Radiological or objective evidence of recurrence or progression on or after the last systemic therapy prior to enrolment.
* CNS metastasis is permitted if asymptomatic and not requiring treatment with steroids and is documented to be non-progressing at study entry
* Presence of measurable or evaluable disease by RECIST 1.1 criteria
* Adequate hematopoietic function: Absolute granulocyte count ≥1,500/mm3, platelet ≥100,000/mm3, hemoglobin ≥ 10g/mm3
* Adequate hepatic function: total bilirubin ≤ 1.5 x upper normal limit (UNL), AST/ALT ≤2.5 x UNL or ≤5 x UNL if presented with hepatic metastasis
* Fasting serum cholesterol ≤ 300mg/dl and fasting triglycerides ≤ 2.5 x UNL
* Adequate renal function: Serum creatinine ≤1.5mg/dL
* Patients should sign a written informed consent before study entry
* Patients with positive HBV-DNA of HBsAg at screening must initiate prophylaxis with appropriate antiviral medication at least one week prior to treatment start

Exclusion Criteria:

* Known active CNS metastasis
* Patients who received prior therapy with gemcitabine
* Patients with only non-measurable lesions other than bone metastasis (e.g. pleural effusion, ascites).
* Patients with more than 3 prior chemotherapy lines for treating metastatic breast cancer.
* Patients who received prior therapy with mTOR inhibitor or PI3K inhibitor
* Known hypersensitivity to mTOR inhibitors, e.g. Sirolimus (rapamycin).
* Radiotherapy within four weeks prior to enrolment, except radiotherapy to the bone for analgesic purpose or for lytic lesions at risk of fracture. Patients must have recovered from radiotherapy toxicities prior to enrolment.
* Patients who have history of cancer other than in situ uterine cervix cancer or nonmelanotic skin cancer
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus
* Active ulceration of upper gastrointestinal tract
* Other concurrent severe and/or uncontrolled conditions (e.g. uncontrolled diabetes mellitus, active untreated or uncontrolled infection, chronic obstructive or chronic restrictive pulmonary disease including dyspnea at rest from any cause) that could cause unacceptable safety risks or compromise compliance with the protocol.
* Patients with a known history of HIV seropositivity. Screening for HIV infection at baseline is not required.
* Significant symptomatic deterioration of lung function. If clinically indicated, pulmonary function tests including measures of predicted lung volumes, DLco, O2 saturation at rest on room air should be considered to exclude restrictive pulmonary disease, pneumonitis or pulmonary infiltrates.
* Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A at enrolment (rifabutin, rifampicin, clarithromycin, ketoconazole, itraconazole, voriconazole, ritonavir, telithromycin) continuously for at least 7 days during any time period in the last 2 weeks prior to enrolment
* Known hypersensitivity to protocol treatment
* Pregnant or breast feeding
* Peripheral neuropathy ≥ grade 2 (NCI CTCAE version 4.0) at randomization
* Patients unwilling to or unable to comply with the protocol

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
The recommended dose of the combination of gemcitabine, cisplatin and RAD001 (everolimus) in patients with metastatic triple-negative breast cancer | up to 1 year
  phase IB part
Efficacy of gemcitabine and cisplatin with or without RAD001 in patients with metastatic triple-negative breast cancer by evaluating progression free survival (PFS) | up to 5 years
  phase II part

SECONDARY OUTCOMES:
The maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of gemcitabine/cisplatin/RAD001 | up to 1 year
  phase Ib part
number of patients with adverse events as a measure of safety and tolerability | up to 5 years
  phase Ib and phase II
objective response rate | up to 1 year
  phase Ib and phase II
Overall survival (OS) | up to 5 years
  phase Ib and phase II
check biomarkers associated with the response of RAD001: angiogenesis, metabolism, immune cells profiles | up to 5 years
  phaseIb and phaseII

CONTACTS AND LOCATIONS:
Overall Officials: In Hae Park, Doctor, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National cancer center, Goyang-si, Gyeonggido, South Korea